CLINICAL TRIAL: NCT04307030
Title: Multi-center Study on Exploration and Application of Artificial Intelligence Technology-Assisted Heart Sound Recognition System in Children's Congenital Heart Disease Screening
Brief Title: Study on AI Recognition System Of Heart Sound In Congenital Heart Disease Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kun Sun, Professor of Department of Pediatric Cardiology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-20-003
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Congenital Heart Disease in Children
Keywords: Congenital Heart Disease; Artificial Intelligence; Heart Sound
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Heart Auscultation; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 0 ~ 18 years old children: Children During Outpatient or Hospitalization
  Interventions: Diagnostic Test: Heart Auscultation and Echocardiography

INTERVENTIONS:
Diagnostic Test: Heart Auscultation and Echocardiography — Heart auscultation will be done by cardiovascular pediatrician and echocardiography by echocardiologist

SUMMARY:
The objective of this study is to establish AI algorithm based on the deep learning to strengthen the ability to classify the heart murmurs of healthy people and different major or other subdivided congenital heart diseases(CHDs) and to evaluate the effectiveness of artificial intelligence technology-assisted heart sound recognition system (referred to as: Heart sound AI recognition system) for multi-center CHD screening.

DETAILED DESCRIPTION:
This is a multi-center cluster cross-sectional study in CHINA. Heart sounds will be collected by auscultation using an electronic stethoscope in children (0 ~ 18 years old) confirmed with or without CHDs by echocardiography during outpatient or hospitalization in 10 pediatric medical centers. Heart sounds will be visualized as phonocardiogram, and feature extraction will be done after classification of normal and abnormal heart sounds and labeling the characteristics of heart murmurs by pediatric cardiovascular specialists. Artificial intelligence algorithm (machine learning, deep learning, etc.) will be trained to build a heart sounds recognition system with the data mentioned above.We will use the receiver operating characteristic (ROC) curve to compare the ability of recognition and classification of abnormal heart sounds between different artificial intelligence algorithm. Taken the results of echocardiography as the gold standard, we will use the evaluation indexes,such as sensitivity, specificity, accuracy, positive predictive value, negative predictive value, etc, to compare the diagnostic capacity of CHD screening between the AI recognition system and human cardiovascular pediatricians. Our target is to use artificial intelligence technology to assist heart auscultation for CHD screening.

ELIGIBILITY:
Inclusion Criteria:

1. 0 ~ 18 years of age, regardless of gender ；
2. Children with or without congenital heart disease confirmed by echocardiography；
3. On the basis of informed consent，willing to cooperate with our group.

Exclusion Criteria:

1. ≥ 18 years of age;
2. Children who can not undergo echocardiography or other related tests;
3. Subjects who refuse to join in, or who are unwilling to cooperate with the provision of diagnostic and therapeutic data for further analysis and research.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric population during outpatient service or hospitalization in ten pediatric medical centers in CHINA
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Receiver operating characteristic (ROC) of sensitivity | July 2020 to December 2021
  ROC of sensitivity in CHD screening by different artificial intelligence algorithm and auscultation

CONTACTS AND LOCATIONS:
Overall Officials: KUN SUN, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (16):
- China (16):
  - Beijing Anzhen Hospital, Beijing
  - Children's Hospital Affiliated to Chongqing Medical University, Chongqing
  - The First Affiliated Hospital of Guangxi Medical University, Guangxi
  - Guangzhou Women and Children's Medical Center, Guangzhou
  - Children's Hospital Affiliated to Zhejiang Medical University, Hangzhou
  - Hunan Children's Hospital, Hunan
  - Shandong Provincial Hospital, Jinan
  - Kunming Children's Hospital, Kunming
  - Lanzhou University Second Hospital, Lanzhou
  - Linyi Hospital for Women and Children, Linyi
  - Children's Hospital of Shanghai, Shanghai
  - Shanghai Children's Medical Center, Shanghai
  - Shiyan Taihe Hospital, Shiyan
  - Children's Hospital of Soochow University, Suzhou
  - The Second Hospital Affiliated to Wenzhou Medical University, Wenzhou
  - Wuhan Children's Hospital, Wuhan

IPD SHARING:
Plan to Share IPD: Undecided